CLINICAL TRIAL: NCT06696625
Title: Transcutaneous Auricular Vagus Nerve Stimulation in Dry Eye: a Randomized Clinical Trial
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Dry Eye
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DED_taVNS_2024
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Disease
Keywords: taVNS; Dry eye; RCT
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS group (Experimental): taVNS device (Elmmedicare, EC100, Shenzhen, China) was used to apply stimulation for patients.
  Stimulation parameters comprised an electrical current of 1 mA at a frequency of 20 Hz, with a waveform width of 1 ms. Repurposed off-the-shelf devices were utilized for this purpose, with the stimulator generating single square-wave pulses lasting 1 ms each. Enhancing conductivity was achieved by wiping the ear with tap water. The electrodes were placed on the cymba conchae and concha around the affected ear, which is the region of rich vagus nerve branch distribution.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation; Drug: 0.1% sodium hyaluronate eye drop
- Control Group (Sham Comparator): taVNS device (Elmmedicare, EC100, Shenzhen, China) was used to apply stimulation for patients.
  Stimulation parameters comprised an electrical current of 1 mA at a frequency of 20 Hz, with a waveform width of 1 ms. Repurposed off-the-shelf devices were utilized for this purpose, with the stimulator generating single square-wave pulses lasting 1 ms each. Enhancing conductivity was achieved by wiping the ear with tap water. The electrodes were placed on the cymba conchae and concha around the affected ear, which is the region of rich vagus nerve branch distribution. Patients in control group were applied using the same stimulator, stimulation parameters and same sessions. However, the electrodes were placed on the antihelix around the affected ear, which is the region of few vagus nerve branch distribution.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation; Drug: 0.1% sodium hyaluronate eye drop

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — taVNS device (Elmmedicare, EC100, Shenzhen, China) was used to apply stimulation for patients.
  Stimulation parameters comprised an electrical current of 1 mA at a frequency of 20 Hz, with a waveform width of 1 ms. Repurposed off-the-shelf devices were utilized for this purpose, with the stimulator generating single square-wave pulses lasting 1 ms each. Enhancing conductivity was achieved by wiping the ear with tap water. The electrodes were placed on the cymba conchae and concha around the affected ear, which is the region of rich vagus nerve branch distribution.
Drug: 0.1% sodium hyaluronate eye drop — Participants received 0.1% sodium hyaluronate eye drop (HYLO COMOD® eye drops, Ursapharm, Ltd., Germany).

SUMMARY:
Objective: To evaluate the effect of transcutaneous auricular vagus nerve stimulation (taVNS) for the patients with dry eye disease.

Methods: The investigators enrolled 256 patients at Beijing Tongren Hospital. Patients completed questionnaires at baseline, 1 month, 3 months, and 6 months. OSDI score, TBUT, Schirmer I, CFS, SF36, DEQ5, and psychological status to evaluate the therapeutic effects. A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and Age <=65.
2. complaint of DED symptoms for 6 months or longer at screening.
3. ocular surface disease index (OSDI) score of 25 or higher.
4. tear film breakup time (TFBUT) of 5 seconds or less.
5. Schirmer I test without anesthesia of 5 mm or more at 5 minutes.
6. tCFS score of 4 or higher.

Exclusion Criteria:

1. History systemic autoimmune diseases and ocular/periocular malignancy.
2. Clinically relevant slitlamp findings or abnormal lid anatomy.
3. Active ocular allergies and active infection.
4. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | Baseline, month 1, 3, and 6
  The Ocular Surface Disease Index (OSDI) includes 12 questions grouped by poor symptoms and visual disturbance (light sensitivity, eyes feel gritty, painful or sore eyes, blurred vision or poor vision); visual function/tasks (problems when reading, driving at night, working on a computer or watching TV); and environmental questions (problems in windy conditions, places/areas with low humidity or areas that are air conditioned). The scores range from 0 to 100. On the basis of the score, the patient's symptoms can be categorized as normal (0-12), mild dry eye (13-22), moderate dry eye (23-32), or severe dry eye (33-100).

SECONDARY OUTCOMES:
TBUT | Baseline, month 1, 3, and 6
  Tear breakup time (TBUT) is a clinical test used to assess for evaporative dry eye disease. To measure TBUT,
  fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed
  under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between
  the last blink and the appearance of the first dry spot in the tear film, as seen in this progression of these slit lamps' photos over time. A TBUT under 10 seconds is considered abnormal.
Schirmer | Baseline, month 1, 3, and 6
  The Schirmer test is objectively used to measure tear secretion without anesthetized. A healthy eye should wet more than 10 mm of the standard filter strip in 5 minutes. The travel rate along the test strip is proportional to the tear production rate.
CFS | Baseline, month 1, 3, and 6
  Corneal Fluorescein Staining (CFS) was measured using the National Eye Institute (NEI) scale, which ranges from 0 (no staining) to 3 (heavy staining) for each of the 5 areas of the cornea (inferior, superior, central, nasal, and temporal).
  The total score ranging from 0 to 15 is the sum of the 5 regions, with higher scores indicating greater symptom severity.
DEQ-5 | Baseline, month 1, 3, and 6
  The 5-Item Dry Eye Questionnaire (DEQ-5) contains five questions regarding the frequency and intensity of eye discomfort, eye dryness and watery eyes in the past month. The score ranges from 0 to 22, a score > 6 suggests dry eye, with higher scores indicating greater symptom severity.
PHQ-9 | Baseline, month 1, 3, and 6
  Depression was assessed with the 9-item Patient Health Questionnaire (PHQ). Patients were classified as having no depression (PHQ score: 0-4), mild (PHQ, score: 5-9), and moderate to severe depression (PHQ score: 10-27). Scores range from 0 to 27, with higher scores indicating greater symptom severity.
SF-36 | Baseline, month 3, 6 and 12
  36-Item Short Form Health Survey (SF36) measures quality of life on the basis of eight dimensions or concepts
  that are frequently used in health studies. These eight dimensions are estimated from eight subscales that examine
  physical functioning (SF36-PF), role functioning-physical (SF36-RP), bodily pain (SF36-BP), general health (SF36-
  GH), vitality (SF36-VT), social functioning (SF36-SF), role functioning-emotional (SF36-RE), mental health (SF36-MH)
  and reported health transition (SF36-HT). Item responses were ranging from 0 (best) to 100 (worst), with higher scores are equivalent to greater severity of better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- China Beijing TongRen Hospital, Capital Medical University Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No